CLINICAL TRIAL: NCT05660837
Title: Online Social Support Program for Physical and Mental Health of Filipino Migrant Domestic Workers in Hong Kong
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hong Kong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Anirban MUKHOPADHYAY, Professor, Hong Kong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HREP-2022-0170
Record Dates: First submitted 2022-11-07; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Healthy Diet; Mental Health Wellness
Keywords: social support; weight management; emotional support; online support groups; eating behavior; mental health; informational support
MeSH Terms: conditions — Feeding Behavior; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The investigators are providing informational and emotional social support (nutrition, mental health, baking classes) through two different communication modalities (online vs. mixed mode) whose effects will be contrasted against each other and a third, control, condition.
  Treatment 1: Mixed-mode social support group Treatment 2: Online social support group Control: No intervention
Who Masked: Outcomes Assessor
Masking Description: Baseline survey, follow-up survey, and anthropometry measurement will be collected through assessor masked to assignment details.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- T1: Mixed mode social support group (Experimental): This group will receive programs in both online and off-line setting. There will be one face-to-face group session to get to know participant's peer group members. After the in-person group meeting, participants will meet in WhatsApp group. In WhatsApp group, facilitator will provide the following program
  Interventions: Behavioral: T1: Mixed mode social support group
- Online social support group (Experimental): This group will receive the same program as mixed mode social support group. The key differences would be delivery of all program components online.
  Interventions: Behavioral: T2: Online mode social support group
- Control (No Intervention): This is the control group.
  Control group will only participate in baseline and follow-up survey

INTERVENTIONS:
Behavioral: T1: Mixed mode social support group — This group will receive programs in both online and off-line setting. There will be one face-to-face group session to get to know participant's peer group members. After the in-person group meeting, participants will meet in WhatsApp group. In WhatsApp group, facilitator will provide the following program
  1. In person get to know your group member activities
  2. Nutrition information through WhatsApp
  3. Tips and advice to maintain good mental health through WhatsApp
  4. Motivational messages through WhatsApp
  5. Reminder through WhatsApp
  6. In-person baking class x 1 session
  Arms: T1: Mixed mode social support group
Behavioral: T2: Online mode social support group — This group will receive the same program as mixed mode social support group. The key differences would be delivery of all program components online.
  1. Online get to know your group member activities
  2. Nutrition information through WhatsApp
  3. Tips and advice to maintain good mental health through WhatsApp
  4. Motivational messages through WhatsApp
  5. Reminder through WhatsApp
  6. Online baking class x 1 session through WhatsApp
  Arms: Online social support group

SUMMARY:
The goal of this study is to test the effect of informational and emotional social support (via nutrition education, mental health support, and/or baking classes) through two different communication modalities (online vs. mixed mode / hybrid) on physical and mental health outcomes

Our research questions are the following.

1. Does an online social support program that provides informational and emotional support improve diet, anthropometry, and mental health?
2. Does a mixed-mode social support program that provides informational, emotional support through both online and face-to-face mode improve diet, anthropometry, and mental health?
3. Is a mixed mode social support program more effective in improving outcomes? Does meeting the group members face-to-face change the dynamics of online communication? If yes, what are the mechanisms? Are there differences in the following outcomes by communication modality?

   1. Online bonding
   2. Group identity
   3. Quality of relationship

DETAILED DESCRIPTION:
Study design: Randomized controlled trial

1. Study description

   Filipino Migrant Domestic workers (MDWs) working in Hong Kong will be eligible to apply. The investigators will advertise in Newspapers and Facebook commonly read by Filipino MDWs in Hong Kong. The investigators will recruit 400 MDWs over two phases and randomly assign them across three arms, T1) mixed-mode social support program; T2) Online social support program; and C) Control. Online social support program will be delivered through WhatsApp group chat. MDWs will self-fill surveys at Caritas office, but surveys will be assisted by survey enumerators as a group.
2. Logistics

   Due to administrative constraints delivering interventions to 400 participants at the same time, the investigators will deliver interventions over two cohorts.

   Cohort 1 (~200 participants)
   * Oct 31st-Dec 18th 2022 Baseline survey
   * Jan 8th-March 18th 2023 Intervention (10 weeks)
   * March 26th -April 16th 2023 Follow-up survey

   Cohort 2 (~200 participants)
   * Feb 5th-March 19th 2023 Baseline survey
   * March 20th-May 27th Intervention (10 weeks)
   * May 28th - June 25th follow-up survey

   Note 1: The investigators will enroll participants until the scheduled date for baseline survey or until the investigators recruit target sample size, whichever comes earlier.

   Note 2: The investigators will keep the intervention design exactly the same for cohort 1 and cohort 2, and will not analyze data until data collection for both cohort 1 and cohort 2 is complete. Cohort 1 and cohort 2 will be analyzed as one sample.
3. Statistical analysis model - Estimation of treatment effect

In this section, the investigators outline the basic estimation approach to measuring the effect of the treatments on various outcomes.

Our basic treatment effects specification estimates the following equation:

y= β₀ + β₁T1 + β₂T2+ β₃X+ ε where y is the outcome of interest.

T1 and T2 are dummy variables equal to 1 if the participant was randomly assigned to the T1 and T2 group, respectively, and 0 otherwise. β₁ and β₂ represent the effect of being assigned to the specific treatment arm. X is a vector of baseline outcome and individual's characteristics including age, marital status, years working as migrant domestic workers, level of education, received food allowance. ε is an error term. The primary outcome variable, y, include nutrition knowledge, perceived social support, healthy diet, stress, anxiety, and depression. To compare the difference between T1 and T2, we will use F-test coefficient of equality.

ELIGIBILITY:
Inclusion Criteria:

* Filipino
* Migrant domestic worker working in Hong Kong

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female will be eligible to participate. Participant eligibility is based on self-representation.
Enrollment: 400 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Nutrition knowledge score (change) | Change from baseline nutrition knowledge at approximately 3-6 months.
  Questions to test nutrition knowledge, survey questionnaire (score range 0-17, higher score means better outcome)
Perceived social support (change) | Change from baseline perceived social support at approximately 3-6 months.
  Participant's perceived social support score, scale adapted from Oslo social support scale (OSSS-3), survey questionnaire, higher score means better outcome.
Healthy diet practices (change) | Change from baseline diet practices at approximately 3-6 months.
  Questions adapted from "starting the conversation (STC)" food frequency instrument, scale range 0-50, higher score means better outcome, survey questionnaire
Stress (change) | Change from baseline mental health at approximately 3-6 months.
  Screen for stress using DASS-21 questionnaire, survey questionnaire (score range (0-42), higher score means worse outcome
Anxiety (change) | Change from baseline mental health at approximately 3-6 months.
  Screen for anxiety using DASS-21 questionnaire, survey questionnaire, score range (0-42), higher score means worse outcome
Depression (change) | Change from baseline mental health at approximately 3-6 months.
  Screen for depression using DASS-21 questionnaire, survey questionnaire, score range (0-42), higher score means worse outcome

SECONDARY OUTCOMES:
Body mass index (change) | Change from baseline BMI at approximately 3-6 months.
  kg/m2, anthropometry measurements
Waist-to-hip ratio (change) | Change from baseline waist-to-hip ratio at approximately 3-6 months.
  waist circumference (cm) /hip circumference (cm), anthropometry measurements
Waist-to-stature ratio (change) | Change from baseline waist-to-stature ratio at approximately 3-6 months.
  Waist circumference (cm)/Height (cm), anthropometry measurements
Self-efficacy (change) | Change from baseline self-efficacy at approximately 3-6 months.
  four questions, General self-efficacy scale (GSE) survey questionnaire, score range 0-30, higher score means better outcome
Group identity | measured at end-line only ( 3-6 months after baseline survey)
  4 questions: 5 point scale (strongly agree to strongly disagree) , survey questionnaire
Online bonding | measured at end-line only (3-6 months after baseline survey)
  10 questions: 5 point scale (strongly agree to strongly disagree), survey questionnaire
Peer pressure | measured at end-line only (3-6 months after baseline survey)
  10 questions: 5 point scale (strongly agree to strongly disagree), survey questionnaire

OTHER OUTCOMES:
Weight (change) | Change from baseline weight at approximately 3-6 months.
  measured in kg
Waist circumference (change) | Change from baseline waist circumference at approximately 3-6 months
  measured in cm
Hip circumference (change) | Change from baseline hip circumference at approximately 3-6 months.
  measured in cm
Depression (change) | Change from baseline at approximately 3-6 months.
  Created dummy variable (moderate or above) from depression score using DASS-21 questionnaire, survey questionnaire
Anxiety (change) | Change from baseline at approximately 3-6 months.
  Created dummy variable (moderate or above) from anxiety score using DASS-21 questionnaire, survey questionnaire
Stress (change) | Change from baseline at approximately 3-6 months.
  Created dummy variable (moderate or above) from stress score using DASS-21 questionnaire, survey questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong University of Science of Technology, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share the study protocol, analysis plan, informed consent form, and study report for up to 5 years after the study is published.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately after the study is accepted for publication, and available for 5 years
Access Criteria: Those who want access will be asked to contact the Principal Investigator via email.